CLINICAL TRIAL: NCT05004610
Title: Hypertonic Lactate After Cardiac Arrest
Acronym: LATTE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SRB2021260
Record Dates: First submitted 2021-07-30; First posted 2021-08-13 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Cardiac Arrest; Ischemia Reperfusion Injury; Anoxic Brain Injury
Keywords: sodium lactate; cerebral metabolism
MeSH Terms: conditions — Heart Arrest; Reperfusion Injury; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard of care (No Intervention): Patients will receive the standard of care infusion (balanced crystalloids)
- treatement group (Experimental): Sodium lactate infusion 15 µmol/Kg/min
  Interventions: Drug: Sodium Lactate Solution

INTERVENTIONS:
Drug: Sodium Lactate Solution — continuous intravenous infusion of molar sodium lactate
  Other Names: Hyperonic sodium lactate
  Arms: treatement group

SUMMARY:
The study is intended to test the hypothesis that sodium lactate infusion after resuscitation from a cardiac arrest will decrease the magnitude of brain damage, as measured by the serum biomarker concentration of NSE.

DETAILED DESCRIPTION:
Background: In resuscitated patients after cardiac arrest, ischemic brain injury and cardiac depression due to the reperfusion injury are accountable for high mortality rate and poor outcome. Hypertonic sodium lactate (HSL) solutions have been proven to be safe in healthy volunteers and they have shown some benefits in patients with traumatic brain injury and those with myocardial ischemia and could decrease the burden of hypoxic lesions in these organs. The aim of this phase II study is to investigate whether HSL administration could reduce organ damage related biomarkers in serum and if the administrations of these solutions is safe and feasible in resuscitated patients after cardiac arrest.

Design: an investigator initiated, randomized, controlled, open label phase II clinical trial to test the safety and efficacy of the infusion of HSL in resuscitated patients after cardiac arrest admitted to the hospital. After resuscitation from CA, comatose patients will be screened for eligibility and randomized to receive either study treatment as HSL 1M infusion for 24h or standard of care.

Expected outcomes: This controlled trial will assess the safety and efficacy of the 1M HSL infusion in a cohort of comatose resuscitated patients after cardiac arrest. The results of this trial may provide useful information for a larger phase III clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Sustained (> 20 minutes) return of spontaneous circulation (ROSC)
* Comatose (GCS < 9)
* Time to ROSC > 15'

Exclusion Criteria:

* Protected categories (Pregnant women)
* Anticipated withdrawal of support within 24 hours
* Traumatic cause of cardiac arrest
* Body weight at admission > 120Kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
serum NSE | 48 hours after randomization
  NSE serum levels

SECONDARY OUTCOMES:
ICU length of stay | trough study completion, on average 30 days
  number of days in the intensive care unit
Mortality | trough study completion before hospital discharge, on average 90 days
  mortality
Neurological outcome | trough study completion, 90 days after randomization
  Neurological outcome measured by Cerebral Performance Category score at 90 days (1-5, 1 meaning better Neurological outcome)
Hospital length of stay | trough study completion, on average 60 days
  Hospital length of stay
Vasopressors equivalent dose | through study completion, during the first 48 hours after resuscitation
  Vasopressors equivalent dose during the first 48 hours after resuscitation
Seizure rate | through study completion before ICU discharge, on average 14 days
  Seizure rate
Changes in cardiac biomarkers | at randomization, 24 hours, 48 hours and 72 hours after randomization
  Troponin I serum levels
Changes in brain biomarkers | at randomization, after 24 hours, 48 hours and 72 hours
  brain biomarkers including nfL and GFAP
Severe adverse events rate | during study drug administration/day 28 or ICU discharge or death
  Serious adverse events rate
Changes in brain metabolism | within 24h after randomization
  Brain metabolism measured by PET-IRM
Changes in brain perfusion | within 24h after randomization
  brain perfusion measured with early perfusion CT scan
Changes in echocardiographic parameters (systolic) | at randomization, at 24 hours and 48 hours after randomization
  Changes systolic cardiac function assessed by echocardiography
Changes in echocardiographic parameters (diastolic) | at randomization, at 24 hours and 48 hours after randomization
  Changes diastolic cardiac function assessed by echocardiography
identification of optimal perfusion pressure | through study completion, on average 30 days
  identification of optimal perfusion pressure with invasive neuromonitoring
identification of optimal cerebral oxygen tension | through study completion, on average 30 days
  identification of optimal cerebral oxygen tension with invasive neuromonitoring

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Annoni, MD, Principal Investigator — Erasme University Hospital
Locations (1):
- Erasme Hospital, Brussels University Hospital (HUB), Brussels, Belgium, Belgium

IPD SHARING:
Plan to Share IPD: No
IPD may be available on reasonable request to other researchers